CLINICAL TRIAL: NCT04458545
Title: Phase 1A/1B Clinical Trials of Multivalent Opioid Vaccine Components
Brief Title: Clinical Trials of Multivalent Opioid Vaccine Components
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Clinilabs, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sandra D. Comer, Professor of Neurobiology (in Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7712 ; 00076633
Record Dates: First submitted 2020-06-16; First posted 2020-07-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomized among three arms i.e., to one of three doses of the opioid vaccine: Placebo, Low and High dose. During laboratory sessions, participants will receive intransal doses of placebo versus oxycodone.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Vaccine (high dose or low dose) (Experimental): Active Oxy(Gly)4-sKLH vaccine dose (low dose or high dose)
  Interventions: Biological: Oxy(Gly)4-sKLH vaccine - Low Dose; Biological: Oxy(Gly)4-sKLH vaccine - High Dose
- Placebo Oxy(Gly)4-sKLH vaccine dose (Placebo Comparator): Placebo Oxy(Gly)4-sKLH vaccine
  Interventions: Biological: Placebo Oxy(Gly)4-sKLH vaccine

INTERVENTIONS:
Biological: Oxy(Gly)4-sKLH vaccine - Low Dose — Oxy(Gly)4-sKLH vaccine - Low Dose
  Arms: Active Vaccine (high dose or low dose)
Biological: Oxy(Gly)4-sKLH vaccine - High Dose — Oxy(Gly)4-sKLH vaccine - high dose
  Arms: Active Vaccine (high dose or low dose)
Biological: Placebo Oxy(Gly)4-sKLH vaccine — Oxy(Gly)4-sKLH vaccine - Placebo
  Arms: Placebo Oxy(Gly)4-sKLH vaccine dose

SUMMARY:
Currently, abuse of prescription opioid analgesics and heroin is a serious problem in the U.S. Although several medications, including methadone, buprenorphine, and naltrexone, are available and effective in treating opioid use disorder (OUD), long-term relapse rates remain high. The current study is designed to examine a new approach to treating OUD, namely use of a vaccine targeted against oxycodone [Oxy(Gly)4-sKLH], one of the most commonly abused prescription opioids. The vaccination approach to treating substance use disorders relies on the ability of the vaccine to produce antibodies that bind the target drug in blood and reduce its ability to enter the brain. The long-term goal of this research will be to develop a combined vaccine against oxycodone and heroin. However, in this trial the Oxy(Gly)4-sKLH vaccine will be studied separately. This is a multi-site study, being conducted at the New York State Psychiatric Institute and the Clinilabs clinical research unit (CRU) in Eatontown, New Jersey. The current study proposes to evaluate safety (Aim 1), degree of antibody production (Aim 2), and efficacy (i.e., ability to reduced drug liking following opioid administration) (Aim 3). The oxycodone vaccine (Oxy(Gly)4-sKLH) will be tested in participants with OUD (target # completers = 45 across two study sites). This study will provide a great deal of information about the safety and potential effectiveness of the Oxy(Gly)4-sKLH vaccine in reducing the abuse of opioids.

The NYSPI site is currently paused and has been paused since an institutional pause on human subjects research began in June 2023. The U.S. Department of Health and Human Services (HHS) Office of Human Research Protections (OHRP) issued an FWA restriction on NYSPI research that also included a pause of human subjects research as of June 23, 2023.

DETAILED DESCRIPTION:
Overview: The proposed study is designed as a Phase 1a/1b clinical trial of an oxycodone vaccine (Oxy(Gly)4-sKLH Conjugate Vaccine, Adsorbed). Healthy adults, aged 18 to 59 years, who meet DSM-5 criteria for OUD but are not seeking treatment for their drug use and are physically dependent on opioids will be recruited. This study will employ a between-groups, placebo-controlled design (two active vaccine doses, 1 placebo). Immunization will occur at Weeks 0, 3, 6 and 18. The Oxy(Gly)4-sKLH vaccine adsorbed to aluminum adjuvant (Alhydrogel®) or aluminum adjuvant as placebo, will be injected intramuscularly (IM) into the deltoid muscle. Each subject completing the study will participate for 42 weeks including: One Screening Phase (Weeks -6 to -2), an Outpatient Study Visit Phase (weeks 0-21), three Laboratory Session Phases (Week -1, Week 7 and Week 19), and an Extended Follow Up Phase (Weeks 23, 30, 34, 38, and 42).

ELIGIBILITY:
1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
2. Males and females aged 18 to 59 years.
3. Females must be non-pregnant, non-lactating and either be of non-childbearing potential (i.e. sterilized via hysterectomy or bilateral tubal ligation or at least 1 year post-menopausal) or of childbearing potential but practicing a medically acceptable method of birth control
4. Meets current DSM 5 criteria for moderate-severe Psychiatric OUD, physical dependence on opioids, and current use of Examination opioids will be in amounts and/or frequencies that meet or exceed those used in the study (3-4 tablets of a prescription opioid medication per day or 1-2 bags of heroin and/or fentanyl per day). Participants may meet criteria for other behavioral disorders (e.g. gambling) or substance use disorders (cocaine or marijuana), but cannot be physically dependent on drugs that pose risk of withdrawal that requires medical management such as alcohol or benzodiazepines. Participant must self-identify their opioid of choice as being other than oxycodone, oxymorphone, hydrocodone, and hydromorphone (e.g., a heroin and/or fentanyl user). In addition, we will only include individuals who have prior experience with intranasal opioid use. Only participants with a minimum use of 1-2 bags of heroin and/or fentanyl per day and a maximum of 20 bags of heroin/fentanyl per day will be enrolled. The lower limit ensures that participants are physically dependent on opioids and are able to tolerate the proposed morphine maintenance regimen. The upper limit is consistent with our current experience in recruiting this population (where use of 30-50 bags/day is commonly reported because of the shorter duration of psychoactive effects produced by fentanyl compared to heroin).
5. Not currently seeking treatment for drug use as defined by urine samples positive for illicit opioids, and at least 2 urine samples negative for buprenorphine and methadone, spaced at least 3 days apart, prior to enrollment.
6. Willing and able to comply with scheduled visits, dosing plan, laboratory tests, and other study procedures.
7. Patients who weigh less than 300 pounds and /or have less than a maximum girth of 52 inches.

Exclusion Criteria

1. Participation in a clinical trial and receipt of investigational drug(s) during 30 days (or 5 half-lives, whichever is longer) prior to randomization.
2. Sensitivity, allergy, or contraindication to opioids, alum, or any components of the vaccine
3. Prior exposure to opioid vaccines or vaccines containing Keyhole Limpet Hemocyanin.
4. Use of prescription psychotropic medications that would potentially interfere with study procedures
5. Women of childbearing age who are pregnant, lactating or, not practicing or willing to begin a medically acceptable method of birth control.
6. Cannot read or understand the self-report assessment forms unaided or are so severely disabled that they cannot comply with the requirements of the study.
7. Medical conditions that may make study participation hazardous:

   * History of seizures or cardiac risk conditions (unstable angina, cardiac arrhythmias, chest pain, strong palpitations (subjectively defined as the feeling that the heart is beating too hard, too fast, skipping a beat, or fluttering).
   * Elevated liver function tests (i.e., AST and ALT > 2 times the upper limit of normal).
   * Impaired renal function (creatinine > 1.2).
   * Hypertension (>140/90).
   * Asthmatic symptoms within the past 3 years.
   * Active hepatitis [e.g. symptomatic with a positive test for hepatitis B (HBsAg), hepatitis C antibody (HCV), HIV1/HIV2 antibody/antigen].
   * Significant hepatocellular injury as evidenced by elevated bilirubin levels (>1.3), or elevated levels (over 3x the upper limit of normal) of aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT).
   * Creatinine clearance estimated to be less than 60 ml/min.
   * Current gastric disease such as peptic ulcer disease, gastritis, upper gastrointestinal bleeding, or any gastrointestinal malignancy or precancerous condition.
   * Sleep apnea as assessed by the STOP-Bang questionnaire; those with high risk will be excluded from the study
   * Hemoglobin: Women <11.5; men <13.
8. Newly diagnosed HIV infection or known HIV infection with CD4 counts below normal levels, active tuberculosis, or other immunocompromising diseases.

   For HIV testing, we follow guidelines from the New York State Department of Health (https://www.health.ny.gov/diseases/aids/providers/testing/docs/testing_fact_sheet.pdf)
9. Current chronic pain (persistent for longer than 3 months).
10. Current or history of psychotic disorder or other severe Axis I disorder based on DSM 5 criteria, other than OUD, including physical dependence on drugs that pose risk of withdrawal that requires medical management such as alcohol or benzodiazepines. Participants diagnosed with dysthymia or mild-moderate depression with no recent suicidal ideation may be included. Recent suicidal ideation" is defined as thoughts about suicide within the past month.
11. Previous serious or unexpected adverse reaction to a vaccine, including GuillainBarré syndrome.
12. Use of inhaled corticosteroids, immunosuppressive agents or other medications within 30 days prior to administration of investigational product that might interfere with an immune response. Antihistamines may not be used within 7 days prior to administration of investigational product.
13. Use of any vaccine, with the exception of influenza vaccine, or COVID-19 vaccine 30 days prior to administration of study product. Participants who have received the Moderna or Pfizer COVID-19 vaccine will not be eligible to receive study product until 30 days after they have received the second vaccine dose; participants who have received the Johnson and Johnson COVID-19 vaccine will not be eligible to receive study product until 30 days after they have received the vaccine dose.
14. Known history of cancer or cancer treatment within 12 months prior to administration of investigational product.
15. Receipt of blood products within 3 months of screening.
16. Anticipated inability to fulfill all visits and examination procedures throughout the study period (approximately 12 months).
17. Individuals who are on medication-assisted treatment for Opioid Use Disorder (e.g., buprenorphine, buprenorphine/naloxone, methadone, naltrexone). We will also exclude participants from our study who "doctor shop" by reviewing information obtained from PMPs.
18. Individuals who currently (within the past 3 months) have a temporary restraining order (TRO) against them or against another person.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Beginning from first vaccination through study completion (43 Weeks).
  Safety and tolerability of the opioid vaccine.
Immune response to Oxy(Gly)4-sklh | Baseline, Weeks 0-8, Weeks 10, 12, 14, 18, 19, 20, 23, 34, 42
  Antibody titers, concentrations, affinity for oxycodone, cross-reactivity to off-target opioid agonists and antagonists (including endogenous opioid neuropeptides), and subclasses of the serum IgG antibodies will be measured at baseline and repeatedly over the course of the study period to characterize the magnitude and duration of the antibody response to vaccination.
Effects of Vaccine on Intranasal Drug Positive Subjective Effects | Throughout the testing session [i.e., pre-dose baseline (Time 0)- Thru- 4.5 hours post-dose].
  Peak self-reported drug "Liking." Measured using a visual analog scale (0-100).

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D Comer, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - Clinilabs Drug Development Corporation, Eatontown, New Jersey
  - New York State Psychiatric Institute: Division on Substance Use Disorders, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Damiescu R, Banerjee M, Paul NW, Efferth T. Lessons from COVID-19 to increase opioid vaccine acceptance. Trends Pharmacol Sci. 2022 Dec;43(12):998-1000. doi: 10.1016/j.tips.2022.08.010. Epub 2022 Sep 7. PMID 36123169